CLINICAL TRIAL: NCT00010998
Title: Yoga: Effect on Attention in Aging & Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Purpose: Treatment
Other Study IDs: P50AT000066-01P3 (NIH); P50AT000066-01 (NIH); NCT00009503 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Yoga
MeSH Terms: conditions — Multiple Sclerosis | interventions — Yoga

INTERVENTIONS:
Procedure: Yoga

SUMMARY:
Changes in visual attention are common among elders and people with multiple sclerosis. The visual attention changes contribute to difficulty with day to day functioning including falls, driving and even finding one's keys on the kitchen counter as well as contributing to deficits in other cognitive domains. Yoga emphasizes the ability to focus attention and there is some evidence that the practice of yoga may improve one's cognitive abilities. Additionally, yoga practice may improve cognitive function through other non-specific means such as improved mood, decreased stress or declines in oxidative injury. We propose a randomized, controlled 6 month phase II trial of yoga in two separate cohorts: healthy elders and subjects with mild multiple sclerosis. We will determine if yoga intervention produces improvements on a broad attentional battery that especially emphasizes attentional control. To further understand the reported beneficial effect of yoga on its practitioners, we will also determine if there is a positive impact on measures directly related to yoga practice (flexibility and balance) as well as mood, quality of life and oxidative injury markers. The yoga intervention consists of a Hatha yoga class meeting twice per week. The class is taught by experienced yoga teachers who are supervised by a nationally known yoga instructor. There are two control groups. An exercise group will have a structured walking program prescribed by a certified Health and Fitness Instructor and Personal Trainer. The program will attempt to match the Hatha yoga class for metabolic demand. The second control group will be assigned to a 6 month waiting list. The outcome measures are assessed at baseline and after the 6 month period. The primary outcome measures are alertness (quantitative EEG and self-rated scale), ability to focus attention (Stroop) and ability to shift attention (extradimensional set shifting task). Secondary attention outcome measures include the ability to sustain attention (decrement in reaction time) and ability to divide attention (Useful Field of View). Other secondary outcome measures include flexibility, balance, mood, quality of life, fatigue (in MS cohort) and decreased markers of lipid, protein, and DNA oxidative injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MS who are mildly impaired with an expanded disability status scale of 0-4.0
* Healthy volunteers

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Dates: Start 1999-09; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Barry S. Oken, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health Sciences University/Neurology, Portland, Oregon, United States